CLINICAL TRIAL: NCT01875107
Title: Insulin Pre-treatment for Steroid-associated Hyperglycemia in Pregnant Diabetic Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Time constraints of primary investigator.
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1301M26861
Record Dates: First submitted 2013-06-03; First posted 2013-06-11 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Hyperglycemia in Pregnant Diabetic Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- insulin pre-treatment (Experimental): insulin pre-treatment of pregnant diabetic patients who receive betamethasone
  Interventions: Drug: insulin pre-treatment

INTERVENTIONS:
Drug: insulin pre-treatment — insulin pre-treatment of pregnant diabetic patients who receive betamethasone

SUMMARY:
Our objective is to assess whether pre-treatment with a fixed dose of insulin, based on weight, given to pregnant patients with gestational or preexisting diabetes receiving betamethasone can provide adequate glycemic control.

Our hypothesis is that pre-treatment with a weight-based calculated insulin dose will help maintain euglycemia for pregnant patients with gestational and preexisting diabetes after steroid administration, and possibly impact length of hospital admission.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women with gestational or pre-existing diabetes admitted to the University of Minnesota
2. Must be 18 years or older
3. Must speak English, Spanish, or Somali
4. Patients must receive steroids for fetal lung maturity as part of their hospital course

Exclusion Criteria:

1. Pregnant women with Type 1 Diabetes, or Type 2 diabetes with evidence of end-organ disease
2. Pregnant women who need to be emergently delivered due to maternal or fetal complications of pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Number of hospital days until euglycemia in pregnant diabetic patients receiving steroids who are pre-treated with insulin. | number of hospital days
  Pregnant diabetic patients admitted to the hospital who receive steroids for fetal lung maturity will have their blood glucose levels checked before and after receiving steroids. Blood glucose levels will be checked fasting and postprandial until the levels are consistently less than 160. This will vary for patients, but will be on average 2 to 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Shelly H Tien,, M.D, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States